CLINICAL TRIAL: NCT03123250
Title: Waterjet Ablation Therapy for Endoscopic Resection of Prostate Tissue II
Acronym: WATERII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0124
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Lower Urinary Tract Symptoms (LUTS); AQUABEAM; Aquablation; Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Aquablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aquablation procedure (Experimental)
  Interventions: Device: Aquablation

INTERVENTIONS:
Device: Aquablation — The procedure is performed with the AquaBeam System. It is designed to utilize a high-velocity sterile saline waterjet as the cutting medium, which is projected through a nozzle positioned within the prostatic urethra. The Aquablation procedure integrates real-time ultrasound imaging with a robotically executed surgeon guided high-velocity waterjet to resect prostate tissue.

SUMMARY:
Single-arm, interventional pivotal clinical trial collecting patient data from use of the AQUABEAM System, a personalized image-guided waterjet resection system that utilizes a high-velocity saline stream to resect and remove prostate tissue in males suffering from Lower Urinary Tract Symptoms (LUTS) due to Benign Prostatic Hyperplasia (BPH) with prostate volumes between 80 mL and 150 mL. The primary endpoints for safety and effectiveness will be measured at 3 months post-treatment. Treated subjects will be followed out to 60 months to collect long-term clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Male age 45-80 years.
* Subject has diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction.
* Subject has an IPSS score greater than or equal to 12.
* Maximum urinary flow rate (Qmax) less than 15mL/s.
* Serum creatinine < 2 mg/dL within 30 days of surgery.
* History of inadequate or failed response, contraindication, or refusal to medical therapy.
* Prostate size ≥ 80 mL and ≤ 150 mL as measured by TRUS.
* Patient is mentally capable and willing to sign a study-specific informed consent form.

Exclusion Criteria:

* BMI ≥ 42.
* Patients unable to stop anticoagulants, antiplatelet agents, or non-steroidal anti-inflammatory agents (NSAIDs, including aspirin greater or equal to 100mg) prior to treatment per standard of care.
* Participants using systemic immune-suppressants including corticosteroids (except inhalants); unable to withhold non-steroidal anti-inflammatory agents (NSAIDs, including aspirin) prior to treatment per standard or care except for low dose aspirin (e.g. less than or equal to 100mg).
* Contraindication to both general and spinal anesthesia.
* Any severe illness that would prevent complete study participation or confound study results.
* History of prostate cancer or current/suspected bladder cancer. Prostate cancer should be ruled out before participation to the satisfaction of the investigator if PSA is above acceptable thresholds.
* History of actively treated bladder cancer within the past two (2) years.
* Clinically significant bladder calculus or bladder diverticulum (e.g., pouch size >20% of full bladder size).
* Active infection, including urinary tract infection or prostatitis.
* Urinary catheter use daily for 90 or more days consecutively.
* Previous urinary tract surgery such as e.g. urinary diversion, artificial urinary sphincter or penile prosthesis.
* Ever been diagnosed with a clinically significant urethral stricture or meatal stenosis, or bladder neck contracture.
* Known damage to external urinary sphincter.
* Has had an open heart surgery, or cardiac arrest < 180 days prior to the date of informed consent.
* Participants using anticholinergics specifically for bladder problems. Use of medications with anticholinergic properties is allowable provided the patient does not have documented adverse urinary side effects from these medications.
* Subject is unwilling to accept a transfusion should one be required.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (13):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Tibor Rubin VA Medical Center, Long Beach, California
  - University of Southern California, Institute of Urology, Los Angeles, California
  - San Diego Clinical Trials, San Diego, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Adult & Pediatrics Urology, Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Toronto-University Health Network, Toronto, Ontario
  - Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhojani N, Bidair M, Kramolowsky E, Desai M, Doumanian L, Zorn KC, Elterman D, Kaufman RP Jr, Eure G, Badlani G, Plante M, Uchio E, Gin G, Paterson R, So A, Roehrborn C, Motola J, Kaplan S, Humphreys M. Aquablation Therapy in Large Prostates (80-150 mL) for Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia: Final WATER II 5-Year Clinical Trial Results. J Urol. 2023 Jul;210(1):143-153. doi: 10.1097/JU.0000000000003483. Epub 2023 Apr 28. PMID 37115632
- [Background] Desai M, Bidair M, Zorn KC, Trainer A, Arther A, Kramolowsky E, Doumanian L, Elterman D, Kaufman RP Jr, Lingeman J, Krambeck A, Eure G, Badlani G, Plante M, Uchio E, Gin G, Goldenberg L, Paterson R, So A, Humphreys M, Roehrborn C, Kaplan S, Motola J, Bhojani N. Aquablation for benign prostatic hyperplasia in large prostates (80-150 mL): 6-month results from the WATER II trial. BJU Int. 2019 Aug;124(2):321-328. doi: 10.1111/bju.14703. Epub 2019 Mar 29. PMID 30734990
- [Background] Desai M, Bidair M, Bhojani N, Trainer A, Arther A, Kramolowsky E, Doumanian L, Elterman D, Kaufman RP Jr, Lingeman J, Krambeck A, Eure G, Badlani G, Plante M, Uchio E, Gin G, Goldenberg L, Paterson R, So A, Humphreys MR, Roehrborn CG, Kaplan S, Motola J, Zorn KC. Aquablation for benign prostatic hyperplasia in large prostates (80-150 cc): 2-year results. Can J Urol. 2020 Apr;27(2):10147-10153. PMID 32333733
- [Background] Desai M, Bidair M, Bhojani N, Trainer A, Arther A, Kramolowsky E, Doumanian L, Elterman D, Kaufman RP Jr, Lingeman J, Krambeck A, Eure G, Badlani G, Plante M, Uchio E, Gin G, Goldenberg L, Paterson R, So A, Humphreys M, Roehrborn C, Kaplan S, Motola J, Zorn KC. WATER II (80-150 mL) procedural outcomes. BJU Int. 2019 Jan;123(1):106-112. doi: 10.1111/bju.14360. Epub 2018 Jun 10. PMID 29694702
- [Background] Bhojani N, Bidair M, Zorn KC, Trainer A, Arther A, Kramolowsky E, Doumanian L, Elterman D, Kaufman RP, Lingeman J, Krambeck A, Eure G, Badlani G, Plante M, Uchio E, Gin G, Goldenberg L, Paterson R, So A, Humphreys M, Kaplan S, Motola J, Desai M, Roehrborn C. Aquablation for Benign Prostatic Hyperplasia in Large Prostates (80-150 cc): 1-Year Results. Urology. 2019 Jul;129:1-7. doi: 10.1016/j.urology.2019.04.029. Epub 2019 May 3. PMID 31059728
- [Derived] Chughtai B, Thomas D. Pooled Aquablation Results for American Men with Lower Urinary Tract Symptoms due to Benign Prostatic Hyperplasia in Large Prostates (60-150 cc). Adv Ther. 2018 Jun;35(6):832-838. doi: 10.1007/s12325-018-0722-0. Epub 2018 Jun 5. PMID 29873008

RESULTS

PARTICIPANT FLOW:
Groups:
- Aquablation Procedure: Aquablation: To utilizes proprietary heat-free high-velocity waterjet technology to resect and remove prostate tissue using the AQUABEAM system, which is a personalized image-guided tissue removal system.
Period: Treatment
Arm/Group | Aquablation Procedure
Started | 101
Completed | 101
Not Completed | 0
Period: 1 Month Follow-Up
Arm/Group | Aquablation Procedure
Started | 101
Completed | 101
Not Completed | 0
Period: 3 Months Follow-Up
Arm/Group | Aquablation Procedure
Started | 99 (2 subjects exited the study since the previous follow-up.)
Completed | 99
Not Completed | 0
Period: 6 Months Follow-Up
Arm/Group | Aquablation Procedure
Started | 100 (Since the previous follow-up, 1 subject who had exited the study was re-enrolled prior to the 6 months follow-up.)
Completed | 100
Not Completed | 0
Period: 12 Months Follow-Up
Arm/Group | Aquablation Procedure
Started | 96 (4 subjects exited the study since the previous follow-up.)
Completed | 96
Not Completed | 0
Period: 24 Months Follow-Up
Arm/Group | Aquablation Procedure
Started | 86 (Since the previous follow-up, 10 subjects did not reconsent to additional long-term follow-ups.)
Completed | 86
Not Completed | 0
Period: 36 Months Follow-Up
Arm/Group | Aquablation Procedure
Started | 82 (4 subjects exited the study since the previous follow-up.)
Completed | 82
Not Completed | 0
Period: 48 Months Follow-Up
Arm/Group | Aquablation Procedure
Started | 66 (Since the previous follow-up, 16 subjects did not reconsent to additional long-term follow-ups.)
Completed | 66
Not Completed | 0
Period: 60 Months Follow Up
Arm/Group | Aquablation Procedure
Started | 62 (4 subjects exited the study since the previous follow-up.)
Completed | 60
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aquablation Procedure
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 5
  Race: Black | 6
  Race: White | 88
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  Canada | 19
  United States | 82
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.2)
Prostate size (TRUS) [Mean (Standard Deviation); unit: cc] — Prostate size as measured through transrectal ultrasound (TRUS).
  cc | 107.4 (22.1)
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: score on a scale] — The objective of the International Prostate Symptom Score (IPSS) is to capture the severity of urinary symptoms related to benign prostatic hyperplasia
  IPSS ranges from 0 to 35. A higher score indicates a worse outcome.
  score on a scale | 23.2 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clavien-Dindo Adverse Events (Percentage of Participants) Through 3 Months Post Treatment
Description: The percentage of subjects with adverse events rated as probably or definitely related to the study procedure classified as Clavien-Dindo Grade 2 or higher or any Grade 1 event resulting in persistent disability (e.g. ejaculatory disorder or erectile dysfunction) evidenced through 3 months post treatment.
Time Frame: 3 months post-treatment
Measure: Number; unit: percentage
Arm/Group | Aquablation Procedure
Number analyzed (Participants) | 101
percentage | 45.5

2. Primary Outcome: Change in Total International Prostate Symptom Score (IPSS) Score at 3 Months as Compared to Baseline
Description: The change in total IPSS score at 3 months as compared to baseline.
  The objective of the International Prostate Symptom Score (IPSS) is to capture the severity of urinary symptoms related to benign prostatic hyperplasia IPSS ranges from 0 to 35. A higher score indicates a worse outcome.
Time Frame: 3 months post-treatment
Population: The number of participants analyzed for this outcome measure consist of the participants who completed the IPSS questionnaire at 3 months post-treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aquablation Procedure
Number analyzed (Participants) | 95
score on a scale | -16.5 [-18.1 to -14.8]

3. Post Hoc Outcome: Change in Total International Prostate Symptom Score (IPSS) Score at 60 Months as Compared to Baseline
Description: The change in total IPSS score at 60 months as compared to baseline
  The objective of the International Prostate Symptom Score (IPSS) is to capture the severity of urinary symptoms related to benign prostatic hyperplasia IPSS ranges from 0 to 35. A higher score indicates a worse outcome.
Time Frame: 60 months post-treatment
Reporting Status: Not Posted, anticipated posting 2023-07

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Aquablation Procedure
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 18/101
Other Adverse Events (participants affected / at risk) | 82/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aquablation Procedure (N=101)
Bleeding (Surgical and medical procedures) | 9 (9)
Cardiac (Cardiac disorders) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Multi-system organ failure (General disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Other (General disorders) | 3 (3)
Scrotal edema (Reproductive system and breast disorders) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aquablation Procedure (N=101)
Bleeding (Surgical and medical procedures) | 8
Dysuria (Renal and urinary disorders) | 12
Ejaculatory dysfunction (Reproductive system and breast disorders) | 23
Pain (General disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 16
Urinary tract infection (Infections and infestations) | 12
Other (General disorders) | 14

LIMITATIONS AND CAVEATS:
The main limitation is that the trial is a single-arm study with a pre-specified performance goal and not randomized against another treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03123250/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT03123250/SAP_001.pdf